CLINICAL TRIAL: NCT02603926
Title: Treatment of Fragile-X Associated Tremor/Ataxia Syndrome (FXTAS) With Allopregnanolone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Randi J. Hagerman, MD (Other)
Responsible Party: Sponsor-Investigator, Randi J. Hagerman, MD, Medical Director, MIND Institute, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 720668
Record Dates: First submitted 2015-11-05; First posted 2015-11-13 (Estimated); Results first posted 2018-12-06 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-11

CONDITIONS: Fragile X-associated Tremor/Ataxia Syndrome
MeSH Terms: conditions — Fragile X Tremor Ataxia Syndrome | interventions — Pregnanolone; brexanolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- Allopregnanolone (Experimental): Subjects will receive an intravenous infusion of Allopregnanolone at escalating doses of 2mg, 4mg, and 6mg once weekly over a three week period. The highest dose tolerated without sedation will be held stable for the remaining weekly infusions, for a total of 12 infusions.
  Interventions: Drug: Allopregnanolone

INTERVENTIONS:
Drug: Allopregnanolone — Allopregnanolone is an endogenous inhibitory pregnane neurosteroid. It is synthesized from progesterone, and is a potent positive allosteric modulator of the action of γ-aminobutyric acid at GABAA receptor. Subjects will receive up to 12 infusions in the study. Subjects will all begin with 2.0 mg dosage. If tolerated, the next infusion will be 4.0 mg, and if that is tolerated, the next infusion will be 6.0 mg. Subject infusions will remain stable at the highest dosage tolerated for the remainder of the study. Each infusion will consist of 2.0 mg, 4.0 mg, or 6.0 mg aliquots of the 0.5 mg/ml allopregnanolone in 6% sulfobutylether-β-cyclodextrin with 0.9% sodium chloride injection solution.
  Other Names: 5α-pregnan-3α-ol-20-one; 3α,5α-tetrahydroprogesterone; brexanolone

SUMMARY:
The purpose of this study is to examine the safety and efficacy of Allopregnanolone as a possible treatment for symptoms of Fragile X-associated Tremor/Ataxia Syndrome (FXTAS).

DETAILED DESCRIPTION:
This study includes a screening visit with several assessments, followed by an open-label medication trial of Allopregnanolone for 12 weeks and an end-point evaluation to assess for changes. Assessments include blood draws for genetic and safety laboratory testing, neurological and physical exam and medical history, cognitive testing, and motor testing.

Study record was updated in October 2018 to include adverse events and outcome measure reporting. Study record was updated in November 2018 in response to requests to (1) specify time frame of reported outcome measures, (2) clarify that the RASS was a safety monitoring tool, not a prespecified outcome measure, and as such will not be reported as an outcome measure, and (3) upload a version of the study protocol and statistical analysis plan with the required title page and statistical analysis plan information.

ELIGIBILITY:
Inclusion Criteria

* Fragile X premutation carrier status (55 to 200 CGG repeats in FMR1),
* Diagnosis of FXTAS including an intention tremor and/or ataxia and/or deficits on the BDS-2 demonstrating executive function deficits.

Exclusion Criteria

* other genetic problems in addition to the premutation
* a history of significant brain trauma
* significant substance abuse
* inability to follow the protocol
* liver or kidney disease
* heart failure
* active cancer
* other serious systemic disease
* current use of phenytoin

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randi J Hagerman, MD, Principal Investigator — UC Davis MIND Institute
Locations (1):
- UC Davis MIND Institute, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited by invitation from the University of California, Davis (UC Davis), MIND Institute's Fragile X Research and Treatment Center.
Groups:
- Allopregnanolone: Subjects will receive and intravenous infusion of Allopregnanolone at escalating doses of 2mg, 4mg, and 6mg once weekly over a three week period. The highest dose tolerated without sedation will be held stable for the remaining weekly infusions, for a total of 12 infusions.
Period: Overall Study
Arm/Group | Allopregnanolone
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Allopregnanolone: Subjects will receive and intravenous infusion of Allopregnanolone at escalating doses of 2mg, 4mg, and 6mg once weekly over a three week period. The highest dose tolerated without sedation will be held stable for the remaining weekly infusions, for a total of 12 infusions.
  Allopregnanolone
Arm/Group | Allopregnanolone
Number analyzed (Participants) | 6
Age, Continuous [Mean (Full Range); unit: years] | 68.3 [57 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: California Verbal Learning Test II (CVLT2) Trial 1-5 Free Recall Total Raw Score
Description: California Verbal Learning Test II (CVLT2) is an assessment measuring working memory. Trials 1-5 measure the total number of words remembered after 5 repeated trials and are summed to generate a raw score (called Trial 1-5 Free Recall Total Raw Score) ranging from 0 to 80, with higher scores reflecting better working memory. Mean and standard deviation for raw score at baseline/pre-treatment and at 14 weeks/post-treatment are presented here.
Time Frame: Baseline/pre-treatment and 14 weeks/post-treatment
Population: Primary outcome measure (CVLT2) was completed for all enrolled subjects.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Allopregnanolone
Number analyzed (Participants) | 6
score on a scale
  Baseline/Pre-Treatment | 34.0 (7.5)
  14 Weeks/Post-Treatment | 33.5 (6.3)

2. Secondary Outcome: Behavioral Dyscontrol Scale - 2 (BDS-2) Total Score
Description: The BDS-2 is a validated 9-item assessment measuring the ability to regulate purposeful, goal-directed activity and to engage in activities of daily living, with focus on motor items. Each of the 9 items is scored on a scale of 0 to 3, resulting in a summed total score ranging from 0 to 27. Higher scores reflect fewer errors and stronger ability to regulate motor activities. Mean and standard deviation for total score at baseline/pre-treatment and at 14 weeks/post-treatment are presented here.
Time Frame: Baseline/pre-treatment and 14 weeks/post-treatment
Population: BDS-2 was completed for all enrolled subjects.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Allopregnanolone
Number analyzed (Participants) | 6
score on a scale
  Baseline/Pre-Treatment | 12.7 (3.1)
  14 Weeks/Post-Treatment | 15.3 (3.8)

3. Secondary Outcome: CATSYS Dot-to-Dot Tremor Intensity (CATSYS DTD TI)
Description: The CATSYS system is a portable device recording various measures of neuromotor control, including tremor. The CATSYS Dot-to-Dot Tremor Intensity (DTD TI) protocol quantifies tremor by having a participant hold a tremor pen as they would an ordinary pen, with the elbow joint bent at a right angle and free of body contact, and the pen positioned approximately 4 inches from the navel. Subjects are instructed to use the pen first to tap the center of two circular stickers, approximately 0.5 inch in diameter, placed on opposite ends of the bottom portion of the computer monitor; then, subjects are instructed to trace a line across the table using the tremor pen. The pen is connected to a computer with sensors that measure tremor intensity (TI) in units of meters per second (m/s). Larger values reflect greater tremor intensity. Mean right-hand and left-hand TI and standard deviation at baseline/pre-treatment and at 14 weeks/post-treatment are reported here.
Time Frame: Baseline/pre-treatment and 14 weeks/post-treatment
Population: CATSYS DTD TI was completed by all subjects.
Measure: Mean (Standard Deviation); unit: meters per second (m/s)
Arm/Group | Allopregnanolone
Number analyzed (Participants) | 6
meters per second (m/s)
  Baseline/Pre-Treatment, Right-Hand | 0.87 (0.49)
  Baseline/Pre-Treatment, Left-Hand | 0.74 (0.29)
  14 Weeks/Post-Treatment, Right-Hand | 0.79 (0.59)
  14 Weeks/Post-Treatment, Left-Hand | 0.65 (0.26)

4. Secondary Outcome: Hippocampal Volume, as Measured by Structural MRI
Description: Patients will undergo structural Magnetic Resonance Imaging (MRI) at baseline/pre-treatment and at 14 weeks/post-treatment. The MRI is interpreted by a trained clinician and hippocampal volume in cubic centimeters is measured and recorded. Larger values reflect greater volumes of the hippocampus, and greater hippocampal volume post-treatment may be indicative of increased neurogenesis. Mean hippocampal volume and standard deviation at baseline/pre-treatment and post-treatment is reported here.
Time Frame: Baseline/pre-treatment and 14 weeks/post-treatment
Population: 1 subject was unable to undergo structural MRI procedure at baseline and post-treatment.
Measure: Mean (Standard Deviation); unit: cubic centimeters
Arm/Group | Allopregnanolone
Number analyzed (Participants) | 5
cubic centimeters
  Baseline/Pre-Treatment | 5.87 (1.00)
  14 Weeks/Post-Treatment | 5.84 (1.18)

ADVERSE EVENTS:
Time Frame: 14 weeks (from baseline to post-treatment).
Description: The Richmond Agitation Sedation Scale (RASS) was administered before, during, and after each infusion; it was not a prespecified outcome measure, rather a safety precaution. Infusions were to be terminated if the score on RASS fellow below -1 (drowsy) during the infusion. Each participant was also required to be accompanied by a chaperone, who drove the participant home from the infusion center and remained with the participant for at least 20 hours thereafter to monitor for adverse effects.
Arm/Group | Allopregnanolone
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
This preliminary trial was conducted to obtain evidence of treatment benefits in a small sample, and thus the study was not powered to detect statistical significance while controlling for multiple comparisons. There was also no placebo group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/26/NCT02603926/Prot_SAP_000.pdf